CLINICAL TRIAL: NCT07327047
Title: How to Place Autogenous Soft Tissue Grafts Ideally for Primary Closure Over Immediately Placed Dental Implants?
Brief Title: Autogenous Soft Tissue Grafts for Primary Closure Over Immediately Placed Dental Implants
Acronym: BFP - FGG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RP.25.05.3
Record Dates: First submitted 2025-12-26; First posted 2026-01-08 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Soft Tissue Augmentation at Dental Implants; Marginal Bone Loss
Keywords: Implantology, Buccal Fat Pad, Immediate Implant, Palatal Gingival Graft, Socket Seal, Soft tissue graft, Posterior Maxilla

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free autogenous soft tissue graft that will be placed without split thickness flaps (Other): Included 10 immediately-placed dental implants with free autogenous soft tissue graft that were placed without split thickness flaps.
  Interventions: Procedure: Free autogenous soft tissue grafts
- Free autogenous soft tissue graft that will be placed within the prepared split thickness flaps (Other): Included 10 immediately-placed dental implants with free autogenous soft tissue graft that were placed within the prepared split thickness flaps
  Interventions: Procedure: Free autogenous soft tissue grafts

INTERVENTIONS:
Procedure: Free autogenous soft tissue grafts — Free autogenous soft tissue grafts (Buccal Pad Fat and Palatal Gingival Graft) that will be placed over immediately-placed dental implants

SUMMARY:
The aim of this interventional study is to evaluate the best method to place the autogenous soft tissue grafts for primary closure over immediately-placed dental implants.

- Primary hypothesis, there is no differences between the two techniques of placement.

DETAILED DESCRIPTION:
The peri-implant mucosa provides protection to the underlying bone via its immune response and protection from apical biofilm migration. An adequate band of attached keratinized mucosa limit early marginal bone loss and improved aesthetic outcomes around implant prostheses. There are several effective socket seal surgery (SSS) techniques to improve the clinical results in the preservation of the alveolar ridge and lessen bone resorption.

Autologous soft tissue grafts still provide the gold standard in gaining keratinized tissue and mucosal thickness compared to autologous substitutes on the market. Simultaneous soft tissue grafts at the time of implant placement can counteract the reduction in ridge width and maintain the ridge architecture regardless of the soft tissue phenotype at the site.

ELIGIBILITY:
Inclusion Criteria:

* Good oral hygiene.
* Medically free from systemic diseases that actually contraindicate implant surgery.
* Patient cooperation.
* The presence of the intact walls of the socket after tooth extraction.

Exclusion Criteria:

* General contraindications for dental and/or surgical treatments.
* Concurrent or previous radiotherapy of head area.
* Smoking.
* Pregnancy.
* Patients refused the procedure.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Marginal Bone Loss | 6 months postoperative
  Marginal Bone Loss around immediately-placed dental implants will be measured in millimeters on cross-sectional view of CBCT

SECONDARY OUTCOMES:
Soft Tissue Healing | At insertion of the prosthetic part (T0) After 2-month post-insertion of the prosthetic part
  Using Pink Esthetic Score

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry - Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No